CLINICAL TRIAL: NCT02245971
Title: A Study on Precutting Methods of Endoscopic Submucosal Dissection for Gastric Neoplasms Located at Lesser Curvature Side of Antrum
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The investigators decided to terminate the study early because there were no patient candidates available for registration in the center.
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2014-0380
Record Dates: First submitted 2014-09-15; First posted 2014-09-22 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Gastric Adenoma and Early Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Whole precutting group (Active Comparator)
  Interventions: Procedure: Whole precutting
- Partial precutting group (Active Comparator)
  Interventions: Procedure: Partial precutting

INTERVENTIONS:
Procedure: Partial precutting — Partial precutting will be performed prior to dissection during the ESD.
  Arms: Partial precutting group
Procedure: Whole precutting — Whole precutting will be performed prior to dissection during the ESD.
  Arms: Whole precutting group

SUMMARY:
Endoscopic submucosal dissection (ESD) is an advanced technique that enables en bloc resection of superficial tumors in the gastrointestinal tract. ESD, however, is a time-consuming procedure that requires a high level of endoscopic skill to achieve a desirable oncologic outcome. Especially, ESD for the lesion which is located in the antrum of lesser curvature side is difficult. Because the antrum of lesser curvature side is dependent position, irrigated water and blood may prevent visual field of ESD.

Generally, whole precutting around the lesion during the ESD is performed prior to dissection. However, it is expected that partial precutting method for the lesion located in the antrum of the lesser curvature may improve the visibility of ESD because it can help us the flap of the lesion evaginated easily. Therefore, we aimed to evaluate the procedure time of ESD for the lesion located in the antrum of the lesser curvature according to the precutting methods (whole precutting vs. partial precutting).

ELIGIBILITY:
Inclusion Criteria:

1. Over 19 years old
2. Patients with gastric adenoma or early gastric cancer

Exclusion Criteria:

1. Patients who has undergone subtotal gastrectomy
2. Patients who has undergone gastrostomy
3. Patients with local recurred gastric adenoma or early gastric cancer

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-07-26 (Actual); Primary Completion 2014-08-12 (Actual); Study Completion 2014-08-12 (Actual)

PRIMARY OUTCOMES:
Procedure time | Within 5 mins after the procedure
  Procedure time for the lesion located in the antrum of lesser curvature according to the precutting methods.

SECONDARY OUTCOMES:
En bloc resection rate | Within 7 days after the procedure
  En bloc resection rate according to the precutting methods.

OTHER OUTCOMES:
complete resection rate | Within 7 days after the procedure
  complete resection rate according to the precutting methods.

CONTACTS AND LOCATIONS:
Locations (1):
- Sevrance hospital, Seoul, South Korea